CLINICAL TRIAL: NCT02914873
Title: SPCG17: Prostate Cancer Active Surveillance Trigger Trial (PCASTT)
Brief Title: SPCG17: Prostate Cancer Active Surveillance Trigger Trial
Acronym: PCASTT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Anna Bill-Axelson, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPCG-17
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; active surveillance; standardised treatment triggers; MRI; randomized
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current clinical practice for active surveillance (Active Comparator): In this arm, patients are monitored according to current clinical practice for active surveillance at the trial centre. Repeat biopsies (and/or other examinations) and curative treatment are performed according to the urologist's judgement.
  Interventions: Procedure: Active surveillance
- Standardized triggers for initiation of treatment with curative intent (Experimental): In this arm, patients are monitored according to a standardized active surveillance protocol with specific triggers for treatment. Repeat biopsies and curative treatment are only initiated if/when specific criteria are fulfilled.
  Interventions: Procedure: Active surveillance

INTERVENTIONS:
Procedure: Active surveillance — Active monitoring of prostate cancer and curative treatment if there are signs of tumor progression.

SUMMARY:
A large proportion of men with prostate cancer are overdiagnosed and overtreated mainly due to PSA testing. Active surveillance (AS) aims to reduce these harms by recommending curative treatment only when and if signs of tumor progression occur. There are however a number of uncertainties in AS, the most important being when to initiate treatment. The investigators are therefore starting a large randomized multicenter trial testing the safety of a standardized active surveillance protocol with specified triggers for repeat biopsies and initiation of curative treatment. The standardized protocol is compared with current practice for active surveillance. The primary aim of the study is to reduce overtreatment and subsequent side effects, without increasing the risk of disease progression or prostate cancer mortality.

DETAILED DESCRIPTION:
STUDY HYPOTHESIS

The study hypothesis is that standardized triggers for initiation of curative treatment of men who are in active surveillance will reduce overtreatment without increasing disease progression and prostate cancer mortality.

STUDY DESIGN

Randomized multi-centre open-label clinical trial

INTERVENTIONS

Computerized randomisation (1:1) within 12 months from diagnosis of prostate cancer, either to active surveillance according to current clinical practice at the trial centre (reference arm), or to a standardised active surveillance protocol applying specific criteria for repeat biopsies and the initiation of curative treatment (experimental arm). Patients are stratified by centre and Gleason score.

Follow-up both groups: PSA every 6 months, clinical examination (with PSA test) annually, and MRI every second year.

Repeat biopsies (reference arm): Current practice

Repeat biopsies (experimental arm), standardised triggers:

1. A systematic repeat biopsy if PSA density increases to > 0.2 ng/ml/cc, and then at every 0.1 ng/ml/cc increase
2. MRI progression in men with previously only Gleason grade 3+3: 5 mm or more increase in size in any dimension of a measurable lesion, increase in PI-RADS score to 3-5, a new lesion with PI-RADS score 3-5, or high or very high suspicion of extra-capsular extension or seminal vesicle invasion
3. MRI progression in men with Gleason grade 3+4: 5 mm or more increase in size in any dimension of a measurable lesion, or a new lesion with PI-RADS score 3-5

Curative treatment (reference arm): Current practice

Curative treatment (experimental arm), standardised triggers:

1. MRI progression in lesions with confirmed Gleason grade 4: increase in PI-RADS score to 4 or 5, or high or very high suspicion of extra-capsular extension or seminal vesicle invasion
2. Pathological progression: Gleason pattern 5, primary Gleason pattern 4 in any core with 5 mm or more cancer, Gleason 3+4 in 3 or more cores or 30% if more than 10 cores are taken, or Gleason 3+4 in 10 mm or more cancer

Patients will be followed continuously until initiation of treatment, the event of metastasis, to a break point where active surveillance is considered terminated and watchful waiting starts, or to death of any cause. For men who discontinue active surveillance, the follow-up and management continue according to standard clinical practice but with annual reporting in the study.

ELIGIBILITY:
Inclusion Criteria:

* Recently (within 12 months) diagnosed adenocarcinoma of the prostate
* Tumor stage less than or equal to T2a, NX, M0
* PSA less than 15 ng/ml, PSA density less than or equal to 0.20 ng/ml/cc
* Gleason pattern 3+3=6 (any number of cores, any cancer involvement)
* Gleason pattern 3+4=7 (less than 3 cores (or less than 30% of cores if more than 10 cores are taken), less than 10 mm cancer in one core)
* Life expectancy more than 10 years with no upper age limit
* Candidate for curative treatment if progression occurs
* Signed written informed consent

Exclusion Criteria:

* none

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2008 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Median 10 years follow-up
  Disease progression is defined as 1) cumulative incidence of PSA relapse after curative treatment or 2) cumulative incidence of androgen deprivation therapy in untreated men still in active surveillance.

SECONDARY OUTCOMES:
Cumulative incidence of pT3 | Median 10 years follow-up
  Occurrence of confirmed pT3 in radical prostatectomy specimens according to the pathology report
Cumulative incidence of metastases | Median 10 years follow-up
  Occurrence of distant metastasis (suspected or confirmed) during follow-up
Cumulative number of treatments with curative intent (mainly radical prostatectomies or local radiotherapy) | Median 10 years follow-up
  Occurrence of radical prostatectomies or local radiotherapy (with or without adjuvant androgen deprivation therapy)
Cumulative incidence of switch to watchful waiting | Median 10 years follow-up
  Occurrence of conversions from active surveillance to watchful waiting during follow-up
Prostate cancer mortality | Median 10 years follow-up
  Prostate cancer-specific mortality at 10 years of follow-up will be analysed, with competing causes of death taken into account.
Quality of life of study participants | Median 10 years follow-up
  Assessed by questionnaire every second year

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bill-Axelson, MD, PhD, Principal Investigator — Uppsala University
Locations (23):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Seinäjoki Central Hospital, Tampere
- Norway (5):
  - Ålesund Regional Hospital, Ålesund
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St Olavs University Hospital, Trondheim
  - Hospital of Vestfold, Tønsberg
- Sweden (8):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Sunderby Regional Hospital, Luleå
  - Örebro University Hospital, Örebro
  - Sundsvall Regional Hospital, Sundsvall
  - Umeå University Hospital, Umeå
  - Akademiska University Hospital, Uppsala
  - Växjö Hospital, Vaxjo
- United Kingdom (6):
  - Bedford Hospital, Bedford
  - Croydon University Hospital, Croydon
  - Epsom and St Helier Hospital, London
  - Guy's Hospital, London
  - Queen Elisabeth Hospital, London
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahlberg MS, Adami HO, Beckmann K, Bertilsson H, Bratt O, Cahill D, Egevad L, Garmo H, Holmberg L, Johansson E, Rannikko A, Van Hemelrijck M, Jaderling F, Wassberg C, Aberg UWN, Bill-Axelson A. PCASTt/SPCG-17-a randomised trial of active surveillance in prostate cancer: rationale and design. BMJ Open. 2019 Aug 22;9(8):e027860. doi: 10.1136/bmjopen-2018-027860. PMID 31444180
- See also: PCASTt/SPCG-17-a randomised trial of active surveillance in prostate cancer: rationale and design — https://bmjopen-bmj-com.ezproxy.its.uu.se/content/9/8/e027860.long

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02914873/SAP_000.pdf